CLINICAL TRIAL: NCT00125970
Title: HVTN Protocol 204 - A Phase II Clinical Trial to Evaluate the Safety and Immunogenicity of a Multiclade HIV-1 DNA Plasmid Vaccine, VRC-HIVDNA016-00-VP, Followed by a Multiclade Recombinant Adenoviral Vector HIV-1 Vaccine Boost, VRCHIVADV014-00-VP, in HIV-1 Uninfected Adult Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 204; 10061 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2005-06-30; First posted 2005-08-02 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 1 (Experimental): DNA HIV vaccine administered at study entry and at Months 1 and 2 and adenoviral vector HIV vaccine administered at Month 6
  Interventions: Biological: VRC-HIVDNA016-00-VP; Biological: VRC-HIVADV014-00-VP
- 2 (Placebo Comparator): DNA HIV vaccine placebo administered at study entry and at Months 1 and 2 and adenoviral vector HIV vaccine placebo administered at Month 6
  Interventions: Biological: VRC-HIVDNA016-00-VP placebo; Biological: VRC-HIVADV014-00-VP placebo

INTERVENTIONS:
Biological: VRC-HIVDNA016-00-VP — 4 mg administered in deltoid
  Other Names: Multiclade HIV-1 DNA Plasmid Vaccine
  Arms: 1
Biological: VRC-HIVADV014-00-VP — 1 x 10^10 PU administered in deltoid
  Other Names: rAD
  Arms: 1
Biological: VRC-HIVDNA016-00-VP placebo — 1 mL administered at study entry and Months 1 and 2
  Other Names: DNA HIV placebo vaccine; Phosphate buffered saline
  Arms: 2
Biological: VRC-HIVADV014-00-VP placebo — 1 mL administered at Month 6
  Other Names: rAD placebo; VRC-DILUENT013-DIL-VP
  Arms: 2

SUMMARY:
The purpose of the study is to determine the safety of and immune response to a DNA HIV vaccine followed by an adenoviral vector HIV vaccine in HIV uninfected adults.

DETAILED DESCRIPTION:
The worldwide HIV/AIDS epidemic may only be controlled through development of a safe and effective vaccine that will prevent HIV infection. DNA vaccines are inexpensive to construct, readily produced in large quantities, and stable for long periods of time. This study will evaluate the safety and immunogenicity of an experimental multiclade HIV vaccine, VRC-HIVDNA016-00-VP, followed by a similarly structured adenovirus-vectored vaccine boost, VRC-HIVADV014-00-VP, in HIV uninfected adults. The DNA plasmids in both the vaccines code for proteins from HIV subtypes A, B, and C, which together represent 90% of new HIV infections in the world. Participants in this study will be recruited in North America, South America, and Africa.

Each volunteer will participate in the study for 36 months. Participants will be randomly assigned to one of two groups. Group 1 participants will receive the DNA HIV vaccine at study entry and at Months 1 and 2. At Month 6, Group 1 participants will receive an injection of the adenoviral vector HIV vaccine. Group 2 participants will receive placebo at study entry and Months 1, 2, and 6. There will be 17 study visits, which will occur at study entry and every 2 weeks thereafter until Day 70; at Month 6 and every 2 weeks thereafter until Day 210; and Months 9.5, 12, 18, 24, 30, and 36. A physical exam, adverse events reporting, HIV and pregnancy prevention counseling, and medication history will occur at each visit. Blood and urine collection will occur at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* Has access to a participating HIV Vaccine Trials Unit (HVTU) and willing to be followed for the duration of the study
* Willing to receive HIV test results
* Good general health
* Willing to use acceptable forms of contraception
* Completed at least 12 years of schooling (South African participants only)

Exclusion Criteria:

* HIV vaccines in prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to first study vaccine administration
* Blood products within 120 days prior to first study vaccine administration
* Immunoglobulin within 60 days prior to first study vaccine administration
* Live attenuated vaccines within 30 days prior to first study vaccine administration
* Investigational research agents within 30 days prior to first study vaccine administration
* Subunit or killed vaccines within 14 days prior to first study vaccine administration
* Current tuberculosis prophylaxis or therapy
* Clinically significant medical condition, abnormal physical exam findings, abnormal laboratory results, or past medical history that may affect current health
* Any medical, psychiatric, or social condition that would interfere with the study. More information about this criterion can be found in the protocol.
* Any job-related responsibility that would interfere with the study
* Serious adverse reaction to vaccines. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Active syphilis infection
* Unstable asthma
* Diabetes mellitus type 1 or 2
* Thyroid disease requiring treatment
* Serious angioedema within the past 3 years
* Uncontrolled hypertension
* Bleeding disorder
* Cancer. If a participant has had surgery to remove the cancer and, in the opinion of the investigator, the cancer is not likely to recur during the study period, the participant is not excluded.
* Seizure disorder
* Asplenia
* Mental illness that would interfere with compliance with the protocol
* Other conditions that, in the judgment of the investigator, would interfere with the study
* Pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2005-09; Primary Completion 2008-02 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Local and systemic adverse reactions | Measured after each injection and for 12 months after the first injection
Unfractionated IFN-γ ELISpot responses to HIV-1 peptide pools as performed by the VRC laboratory | Measured at Day 196
Unfractionated IFN-γ ELISpot responses to HIV-1 peptide pools as performed by the FHCRC laboratory | Measured at Day 210
CD4 and CD8 T cell responses to HIV-1 peptide pools as measured by flow cytometry-based intracellular cytokine staining (ICS) assay as performed by the VRC laboratory | Measured at Day 196
CD4 and CD8 T cell responses to HIV-1 peptide pools as measured by flow cytometry-based ICS assay as performed by the FHCRC laboratory | Measured at Day 210

SECONDARY OUTCOMES:
Humoral immune response to HIV-1 as measured by neutralizing antibody and binding assays | Measured through Month 36
Unfractionated IFN-γ ELISpot responses to HIV-1 as performed by the FHCRC or the VRC laboratories | Measured at Days 70, 210, and 364
CD4 and CD8 T cell responses to HIV-1 as measured by flow cytometry-based ICS assay as performed by the FHCRC or the VRC laboratories | Measured at Days 70, 210, and 364
Vaccine-induced HIV-specific T cell responses to individual peptide pools as measured by IFN-γ ELISpot and ICS as performed by the FHCRC or the VRC laboratories | Measured through Month 36
Cross-clade cellular immune responses to HIV-1 Gag-Pol-Nef peptides from clades A and C as assessed by IFN-γ ELISpot and ICS assays as performed by the FHCRC or the VRC laboratories | Measured through Month 36

CONTACTS AND LOCATIONS:
Overall Officials: Michael Keefer, MD, Study Chair — University of Rochester; Gavin Churchyard, MBBCh, FCP, MMed, PhD, Study Chair — Aurum Health Research Limited
Locations (12):
- United States (5):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - Project Brave HIV Vaccine CRS, Baltimore, Maryland
  - Brigham and Women's Hosp. CRS, Boston, Massachusetts
  - Miriam Hospital's HVTU, Providence, Rhode Island
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
- Brazil (2):
  - Projeto Praca Onze/Hesfa Crs, Rio de Janeiro
  - Sao Paulo HVTU - CRT DST/AIDS CRS, São Paulo
- Les Centres GHESKIO CRS, Port-au-Prince, Haiti
- Epidemiology Research & Training Unit Jamaica MOH CRS, Kingston, Jamaica
- South Africa (3):
  - Soweto HVTN CRS, Johannesburg, Gauteng
  - Emavundleni Desmond Tutu HIV Centre CRS, Cape Town
  - CAPRISA Aurum CRS, Klerksdorp

REFERENCES:
- [Background] Esparza J, Osmanov S. HIV vaccines: a global perspective. Curr Mol Med. 2003 May;3(3):183-93. doi: 10.2174/1566524033479825. PMID 12699356
- [Background] Gaschen B, Taylor J, Yusim K, Foley B, Gao F, Lang D, Novitsky V, Haynes B, Hahn BH, Bhattacharya T, Korber B. Diversity considerations in HIV-1 vaccine selection. Science. 2002 Jun 28;296(5577):2354-60. doi: 10.1126/science.1070441. PMID 12089434
- [Background] Moore JP, Parren PW, Burton DR. Genetic subtypes, humoral immunity, and human immunodeficiency virus type 1 vaccine development. J Virol. 2001 Jul;75(13):5721-9. doi: 10.1128/JVI.75.13.5721-5729.2001. No abstract available. PMID 11390574
- [Background] Stratov I, DeRose R, Purcell DF, Kent SJ. Vaccines and vaccine strategies against HIV. Curr Drug Targets. 2004 Jan;5(1):71-88. doi: 10.2174/1389450043490686. PMID 14738219
- [Derived] Fischinger S, Cizmeci D, Deng D, Grant SP, Frahm N, McElrath J, Fuchs J, Bart PA, Pantaleo G, Keefer M, O Hahn W, Rouphael N, Churchyard G, Moodie Z, Donastorg Y, Streeck H, Alter G. Sequence and vector shapes vaccine induced antibody effector functions in HIV vaccine trials. PLoS Pathog. 2021 Nov 29;17(11):e1010016. doi: 10.1371/journal.ppat.1010016. eCollection 2021 Nov. PMID 34843602
- [Derived] Jin X, Morgan C, Yu X, DeRosa S, Tomaras GD, Montefiori DC, Kublin J, Corey L, Keefer MC; NIAID HIV Vaccine Trials Network. Multiple factors affect immunogenicity of DNA plasmid HIV vaccines in human clinical trials. Vaccine. 2015 May 11;33(20):2347-53. doi: 10.1016/j.vaccine.2015.03.036. Epub 2015 Mar 25. PMID 25820067
- [Derived] Churchyard GJ, Morgan C, Adams E, Hural J, Graham BS, Moodie Z, Grove D, Gray G, Bekker LG, McElrath MJ, Tomaras GD, Goepfert P, Kalams S, Baden LR, Lally M, Dolin R, Blattner W, Kalichman A, Figueroa JP, Pape J, Schechter M, Defawe O, De Rosa SC, Montefiori DC, Nabel GJ, Corey L, Keefer MC; NIAID HIV Vaccine Trials Network. A phase IIA randomized clinical trial of a multiclade HIV-1 DNA prime followed by a multiclade rAd5 HIV-1 vaccine boost in healthy adults (HVTN204). PLoS One. 2011;6(8):e21225. doi: 10.1371/journal.pone.0021225. Epub 2011 Aug 3. PMID 21857901